CLINICAL TRIAL: NCT01560533
Title: Representation of the Body and Treatment of Peritoneal Cancer by Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) - A Collaborative Approach Between Professionals of Health / Patients / Researchers
Brief Title: Representation of the Body for Patients With Cancer
Acronym: CORCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010.640
Record Dates: First submitted 2011-12-12; First posted 2012-03-22 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-01

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated by HIPEC (Other): Patients treated by HIPEC for peritoneal cancer
  Interventions: Behavioral: Interviews
- Standard chemiotherapy (Other): Patients treated by standard chemiotherapy for peritoneal cancer
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — Interviews will be done with patients

SUMMARY:
The project aims to understand better how patients live the event of cancer and live its consequences on their bodily representations. In the study, the dynamic of the body image is not restricted to appearance but include sensations and visions of the inner body, what explains the choice of peritoneal cancer, and the treatment by cytoreductive surgery and HIPEC.

The three objectives of the study are:

* identifying the impact of the representations of the treated body on the psychological strategies to cope with the disease, the bodily changes and the prospects of life;
* making explicit the positive or negative impacts of these representations on the relationship between patients and health professionals (easing factors, misunderstandings, negotiations, etc.);
* associating the health professionals with the study in its course and evaluation in order to elaborate a methodological collaborative approach between patients, health professionals and researchers in social sciences.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to treatment of cancer by cytoreductive surgery and HIPEC
* Primary (pseudomyxoma, mesothelioma) and secondary (colorectal, gastric, ovarian) peritoneal cancer
* Free consent
* Male or Female
* Age > 18 years
* Affiliate to social security

Exclusion Criteria:

* Age < 18 years, no french speaking
* Cerebrals metastasis
* Psychiatrics diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Body representations | 3 months
  Comprehensive knowledge concerning the way the patients are living cancer event, treatment, changes in their body representations and conceptions of their lives.
  This qualitative study do not include outcome measures. Its purpose is restricted to the meanings

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GLEHEN, Pr, Principal Investigator — Hospices Civiles de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Result] Durif-Bruckert C, Guilloux R, Guioux A, Lasserre E, Goffette J, Regnier V. [Qualitative and collaborative research with cancer patients. Experience narratives of treatments for peritoneal carcinomatosis]. Bull Cancer. 2016 Feb;103(2):148-53. doi: 10.1016/j.bulcan.2015.10.015. Epub 2015 Dec 8. French. PMID 26681640